CLINICAL TRIAL: NCT06966128
Title: The Effect of Transcranial Direct Current Stimulation on Cerebral Blood Flow in Patients With Multiple Sclerosis
Brief Title: Transcranial Electrical Stimulation in Multiple Sclerosis
Acronym: TEMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 24378_TEMS; FWOAL1107 (Other Grant/Funding Number: Fund for Scientific Research, Flanders, Belgium)
Record Dates: First submitted 2025-01-06; First posted 2025-05-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cerebral hemodynamics; Cerebral circulation; Cerebral hypoperfusion; Transcranial Direct Current Stimulation; Electrical stimulation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham-first tDCS (Other): The sham-first group will receive: Sham stimulation in visit 1, Active stimulation in visit 2
  Interventions: Device: transcranial Direct Current Stimulation
- Active-first tDCS (Other): The active-first group will receive: Active stimulation in visit 1, Sham stimulation in visit 2
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — Stimulation intensity: Variable (between 1 mA and 2 mA), Electrode placement: Dorsolateral prefrontal cortex, Duration: 10 minutes

SUMMARY:
First the investigators will examine if the blood flow in the brain is different in patients with Multiple Sclerosis compared to healthy volunteers.

HOW?

- The blood flow of the subjects is imaged by use of a special MRI-technique.

Secondly, the investigators will examine if the blood flow can determine disease progression.

HOW? - Multiple Sclerosis patients are asked for a follow-up visit after two years.

The main goal is to understand the effect of transcranial Direct Current Stimulation (tDCS) on the cerebral blood flow.

* Does tDCS result in a different blood flow, in which brain regions?
* Is there a difference between healthy volunteers and Multiple Sclerosis patients?

HOW?

- Participants get two session of tDCS. Before, during and after stimulation MRI scans are performed.

DETAILED DESCRIPTION:
Comparison of CBF between healthy volunteers and MS patients:

- Arterial spin labelling (ASL) is used to investigate cerebral blood flow in patients with MS and healthy volunteers.

The effect of transcranial direct current stimulation (tDCS) on cerebral blood flow:

* ASL scans are performed before-, during-, and after tDCS
* Each subject will receive active and sham tDCS (seperated by at least two days) (cross-over design).

Follow-up visit:

* After two years, patients with MS are re-invited.
* This visit will include a new neuropsychological evaluation, blood sampling and additional brain scans.

ELIGIBILITY:
Inclusion criteria - MS patient

* EDSS ≥ 2 and EDSS ≤ 6.5
* Age ≥ 18

Exclusion criteria - MS patient

* EDSS > 6.5
* Incompatibility with MRI
* Relapse within three months before the study and its use of corticosteroids
* Disabling concomitant neuropsychiatric diseases
* Chance of pregnancy, breastfeeding
* Contraindications to tDCS

Inclusion criteria - Healthy Volunteer

• Age ≥ 18

Exclusion criteria - Healthy Volunteer

* Incompatibility with MRI
* Disabling concomitant neuropsychiatric diseases
* Chance of pregnancy, breastfeeding
* Contraindications to tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow (CBF) | Visit 1 (baseline), visit 2 (+-1 week after visit 1), visit 3 (2 years after visit 1)
  Measure of brain perfusion.
  CBF is measured at baseline and after two years. Additionally, the investigators will measure CBF before-, during-, and after tDCS.

SECONDARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) | Baseline and after 2 years
  Measure of information processing speed
California Verbal Learning Test (CVLT-II) | Baseline and after 2 years
  Measure of verbal memory
Controlled Oral Word Association Test (COWAT) | Baseline and after 2 years
  Measure of verbal fluency
Brief visuospatial Memory Test (BVMT-R) | Baseline and after 2 years
  Measure of spatial memory
Fatigue Scale for Motor and Cognitive Function (FSMC) | Baseline and after 2 years
  Measure of fatigue
Beck's depression inventory (BDI) | Baseline and after 2 years
  Measure of depression
MRI T1 scan | Baseline and after 2 years
  Cortical volume, volumes of white matter and deep grey matter
MRI T2 FLAIR scan | Baseline and after 2 years
  Lesion load, lesion volume

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University hospital of Brussels, Brussels
  - National MS Center Melsbroek, Melsbroek

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data. As we collect personal data on people with multiple sclerosis, we share data on request and after signing a data sharing agreement between both parties. This ensures proper usage and interpretation of the results.